CLINICAL TRIAL: NCT04189822
Title: Hearts in Rhythm Organization (HiRO)National Registry and Bio Bank: Improving Detection and Treatment of Inherited Heart Rhythm Disorders to Prevent Sudden Death
Brief Title: Hearts in Rhythm Organization (HiRO)National Registry and Bio Bank
Acronym: HiRO
Status: Enrolling by invitation | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Andrew Krahn, Professor, University of British Columbia
Other Study IDs: H19-01358
Record Dates: First submitted 2019-11-18; First posted 2019-12-06 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Sudden Cardiac Arrest; Sudden Arrhythmic Death Syndrome; Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC); Long QT Syndrome (LQTS); Hypertrophic Cardiomyopathy (HCM); Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT)
Keywords: Sudden Cardiac Arrest; Inherited Heart Rhythm Conditions; Cardiogenetics
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmogenic Right Ventricular Dysplasia; Long QT Syndrome; Cardiomyopathy, Hypertrophic; Polymorphic Catecholaminergic Ventricular Tachycardia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood Samples drawn:
  1 X 9 ml EDTA
  1 X 10 ml redtop serum tub
  Saliva may be collected as an alternative to blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hearts in Rhythm Organization (HiRO) is a national network of Canadian researchers/clinicians, working towards a better understanding of the rare genetic causes of sudden cardiac death (SCD).

Canadian adult and pediatric electrophysiology centres across Canada work together to gather data and bio sample in a national data registry and bio bank hoping to improve the detection and treatment of inherited heart rhythm disorders to prevent sudden death.

DETAILED DESCRIPTION:
Led by clinical researchers, HiRO is focused on identifying phenotype-genotype correlations. HiRO has defined the investigation pathway for patients with possible genetically mediated cardiac arrest, and has had major impact on our understanding of familial sudden death. However, because many of the Canadian clinics lack a system of care or embedded research, it is difficult to translate novel discoveries to improved care. This current protocol provides a system wide mechanism to allow the national investigator group to work together more efficiently to ensure the inclusion of all Canadians affected by the inherited causes of SCD to help ensure standardized quality care for this population in all provinces with embedded opportunity for all individuals to participate in research.

Background:

Inherited Heart rhythm disorders include arrhythmogenic right ventricular cardiomyopathy (ARVC), Brugada Syndrome, Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT) and Long QT Syndrome (LQTS). They affect one in 200 Canadians and can result in tragic sudden cardiac death (SCD), reduced quality of life and productivity, and high health care expenditure. SCD kills 30,000 Canadians/year. Importantly, clinical screening for at-risk individuals has tremendous potential for timely monitoring and treatment. Treatment typically involves lifestyle modifications, such as avoidance of strenuous exercise, drugs that may worsen the phenotype or medical therapy with beta-blockers or quinidine which can provide substantial protection from SCD. Patients who have cardiac events while on medical therapy, have suffered an unexplained cardiac arrest (UCA), or are deemed sufficiently high risk are offered an implantable cardioverter defibrillator (ICD). ICD therapy provides protection however, it is commonly associated with life-long device related complications.

Patients reviewed in partnering HiRO, Inherited Heart Rhythm Clinics will be invited to participate in the registry.

Optional bio bank participation:

Participants will be invited to provide a blood or saliva sample for storage for future research.Central bio banking for all national bio banks will be available at the lead centre in Vancouver in the James Hogg lab at St. Paul's Hospital in Vancouver BC

Data Collection:

Clinical data will be collected from willing/consented registry participants. Their healthcare information will be coded in compliance with Tri Council Policy Statement criteria: direct identifiers will be removed and replaced with a unique study code that does not use personal information such as the participant's birth day (month and year will be included), health number, social insurance number or name/initials. The coded data will be transferred into the research database.

The master list of registry participants with their study identifiers will be kept separately from the research database. This master list will be stored in an encrypted file within the research office of each site investigators under their supervision. Only the site investigators and their local research staff will have access to this list. The inherited nature of these conditions makes the master list an important and very sensitive document. It will be very important that this list is maintained so that participants may be contacted and informed of any new findings the research may reveal that may affect themselves and their family members.

All medical information pertaining to the cardiac history of inherited arrhythmia patients will be collected. This may include:

* Clinical information
* All diagnostic test results Genetic screening results
* Pedigree
* Medications
* Treatments
* Race Participants will continue to have their data collected for the research database throughout the entirety of the study. Participants will be able to decline further participation in the registry at any time.

Follow-up:

Participants are reassessed as part of clinical care every 3 years in person, collecting the same data as at baseline; this is a repeat phenotyping cycle and reflects standard clinical practice in Canada in the adult IHR population.

Research Data system:

The data base will be maintained by the HiRO research coordinating centre in Vancouver BC. The database will be hosted on the Amazon Virtual Private Network. This network is in compliance with National Canadian/Provincial PIPEDA privacy guidelines. Data will be entered directly into the e-CRFs for electronic submission to a password protected internet-based server located in Montreal Quebec Canada.

Individual participant medical information obtained as a result of this registry is considered confidential and disclosure to third parties is prohibited except for the following reason: relevant medical information may be given to the participant's personal physician or to other appropriate medical personnel responsible for the participant's welfare.

Bio Bank:

Biological (blood or saliva) samples will be coded in compliance with Tri Council Policy Statement criteria: direct identifiers will be removed and replaced with a unique study code that does not use personal information such as the participant's birth date, health care number, social insurance number or name/initials. The coded samples will be linked to the master list kept securely in the research office of the individual investigators. Each sub site investigator and their local research staff will have access to the master list of their local patients only. These master lists will not be shared amongst the investigators.

Blood Samples drawn:

1 X 9 ml EDTA

1 X 10 ml redtop serum tube

Saliva sample: cheek swab

Samples for bio banking will be managed by the coordinating centre in Vancouver British Columbia stored long-term in the James Hogg Research Centre (JHRC) Bio Bank at St. Paul's Hospital in Vancouver for future research.

Oversight

HiRO Research Steering Committee (HRSC) for the National HiRO research registry and bio bank:

The HRSC will be responsible for the design, execution, analysis, and reporting of the study, and will assign appropriate responsibilities to the other study committees. The HRSC will monitor study progress, execution and management. This committee will be responsible for the integrity of the study data and samples. They will also be responsible for reviewing and approving sub study proposals, for use of the registry data and bio samples.

The committee members are:

Dr. Jason Roberts (London Health Sciences) Dr. Andrew Krahn (University of BC/Vancouver) Dr. Rafik Tadros (Montreal Heart Institute) Julia Cadrin -Tourginy (Montreal Heart Institute) Dr. Ciorsti MacIntyre (Dalhousie/Halifax) Dr. Christian Steinberg (Laval/Quebec) Dr. Martin Gardner (Dalhousie/Halifax) Dr. Martin Green (Ottawa Heart Centre)

National HiRO Patient/Public Partners when appropriate will review and advise on projects to provide the patient perspective of the research questions and will propose patient oriented research projects.

Database/bio bank access and Oversight:

The HRSC will have ultimate responsibility for the database. All Investigators on the HRSC listed in this protocol will have equal access to the de-identified data once they have signed the HRSC charter (* see attachment #3*). The HRC investigators will be responsible for annual reviews of data collection, to ensure completeness and accuracy

Proposed sub- studies involve an established proposal submission form, discussion, formal presentation to the HRSC for approval, and a robust lab manual that defines sample access, handling, analysis and reporting.

Only aggregate coded data would be released for these purposes. These data/specimens may be used by a variety of sources. It is anticipated that there may be requests to pool de-identified data/specimens with data/specimens from other international registries/banks in order to answer investigator initiated questions about patient selection, rare events, and long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All Canadian patients referred for cardiac investigations related to inherited heart rhythm (IHR) conditions will be invited to participate if they meet the following criteria:

  * They understand the registry/bio bank purpose, potential risks and willingly sign consent
  * Recognized genetic syndromes; Long QT syndrome (LQT), Short QT Syndrome (SQT), catecholaminergic polymorphic ventricular tachycardia (CPVT), Brugada (BrS), Arrhythmogenic Right Ventricular Cardiomyopathy (ARVC), Familial Cardiac Conduction Disease (FCCD).
  * Deceased cases of SCD, suspicious for an inherited heart rhythm condition. Included with signed consent from next of kin (NOK).
  * IHR patients referred for risk of SCD enrolled (includes first degree and second degree relatives) SCD syndromes seen in heart rhythm clinics; Unexplained cardiac arrest (UCA), Early Repolarization (ER), Idiopathic Ventricular Fibrillation (IVF), Short Coupled IVF (SCIF), Polymorphic Ventricular Tachycardia Not Otherwise Diagnosed (PMVT, NYD), Sudden Arrhythmic Death Syndromes (SADS) that are SCD cases with negative autopsy results.
  * Mendelian cardiomyopathies (hypertrophic cardiomyopathy (HCM), Mendelian Dilated Cardiomyopathy (DCM) including Lamin and Phosopholambin (LMNA, & PLN), and Left Ventricular Non -Compaction (LVNC).

    **Must have either a probable or definite clinical diagnosis, first degree relative (FDR) with a known diagnosis, gene carrier (disease causing or likely disease causing by American College of Medical Genetics (ACMG 2015), or may be second degree relative (SDR) with inability to screen intervening relative
  * Carriers of a pathogenic or likely-pathogenic variant for an inherited arrhythmia or cardiomyopathy related gene, not otherwise fitting inherited or cardiomyopathy diagnostic criteria

Exclusion:

Patients referred for cardiac investigations related to inherited heart rhythm conditions will be excluded from participating if they meet the following criteria:

* Unwilling or are unable to provide informed consent
* Known sarcoidosis
* Mitral valve Prolapse unless unexplained cardiac arrest or syncope with documented PMVT
* Heart Failure/Non-Familial Dilated Cardiomyopathy DCM without a positive family history of affected FDRs or SDRs
* Aortopathies including Marfan Syndrome, Ehlers Danlos, Familial Thoracic Aortic Aneurysm and Dissection
* Neuromuscular disease
* Familial hypercholesterolemia

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The registry will include all willing participants seen as patients in the HiRO network that are evaluated for familial risk of sudden death. The registry will include, inheritable heart rhythm conditions including but not restricted to; Brugada Syndrome, Long QT syndrome, hypertrophic cardiomyopathy (HCM), catecholaminergic polymorphic ventricular tachycardia (CPVT), and arrhythmogenic right ventricular cardiomyopathy (ARVC) and uncommon variants of ARVC that are listed fully in the inclusion criteria section of this protocol as well as first degree family members.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Create a Canadian Research Data base and Bio bank for those affected by inherited heart rhythm conditions. | November 2019 - June 2025
  To build a data registry and bio bank of 10,000.00 inherited heart rhythm cases

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia/St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellor G, Laksman ZWM, Tadros R, Roberts JD, Gerull B, Simpson CS, Klein GJ, Champagne J, Talajic M, Gardner M, Steinberg C, Arbour L, Birnie DH, Angaran P, Leather R, Sanatani S, Chauhan VS, Seifer C, Healey JS, Krahn AD. Genetic Testing in the Evaluation of Unexplained Cardiac Arrest: From the CASPER (Cardiac Arrest Survivors With Preserved Ejection Fraction Registry). Circ Cardiovasc Genet. 2017 Jun;10(3):e001686. doi: 10.1161/CIRCGENETICS.116.001686. PMID 28600387
- [Background] Krahn AD, Healey JS, Chauhan V, Birnie DH, Simpson CS, Champagne J, Gardner M, Sanatani S, Exner DV, Klein GJ, Yee R, Skanes AC, Gula LJ, Gollob MH. Systematic assessment of patients with unexplained cardiac arrest: Cardiac Arrest Survivors With Preserved Ejection Fraction Registry (CASPER). Circulation. 2009 Jul 28;120(4):278-85. doi: 10.1161/CIRCULATIONAHA.109.853143. Epub 2009 Jul 13. PMID 19597050
- [Background] Herman AR, Cheung C, Gerull B, Simpson CS, Birnie DH, Klein GJ, Champagne J, Healey JS, Gibbs K, Talajic M, Gardner M, Bennett MT, Steinberg C, Janzen M, Gollob MH, Angaran P, Yee R, Leather R, Chakrabarti S, Sanatani S, Chauhan VS, Krahn AD. Outcome of Apparently Unexplained Cardiac Arrest: Results From Investigation and Follow-Up of the Prospective Cardiac Arrest Survivors With Preserved Ejection Fraction Registry. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003619. doi: 10.1161/CIRCEP.115.003619. PMID 26783233
- See also: HiRO website — http://heartsinrhythm.ca